CLINICAL TRIAL: NCT03918564
Title: An Investigative, Prospective, Non-randomized, Multi-center Study to Assess the Safety and Effectiveness of a Novel Gastric Restrictive Device, Call the ReShape Vest™, in People Who Are Obese.
Brief Title: ReShape Vest™ for the Treatment of Obesity (Europe)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDURE II
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Weight Loss
Keywords: Weightloss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Laparoscopic Gastric Vest (LGV) — The Laparoscopic Gastric Vest (LGV), branded the ReShape Vest™, is a long-term, silastic, implantable system that is placed around the stomach to encompass the gastroesophageal junction to the Incisura Angularis.
  The main materials used to make the LGV is Implant Grade Silicone (95%) and Barium Sulfate (5%).
  The LGV is indicated for weight reduction for obese people with a Body Mass Index (BMI) between ≥35 kg/m2 and ≤55 kg/m2. It is indicated for use in adult patients (≥22 to ≤65 years) who have failed one or more conservative weight reduction alternative(s), such as supervised diet, exercise, and behavior modification program(s).
  Other Names: ReShape Vest™

SUMMARY:
To assess the safety and effectiveness of the LGV in treating obese subjects with a BMI of 35 kg/m2 to 55 kg/m2 who have failed one or more conservative weight-reduction alternative(s), such as supervised diet, exercise, and behavior modification program(s).

ELIGIBILITY:
Inclusion Criteria:

* Obesity class II and III (Body mass index (BMI) ≥ 35 kg/m2 to ≤55 kg/m2);
* Failed one or more conservative weight-reduction alternative(s), such as supervised diet, exercise, and behavior modification program(s) within the last five years;
* Able to comprehend, follow and give signed informed consent;
* Reside within a reasonable distance from the Investigator's treating office and able and willing to travel to the Investigator's office to complete all routine follow-up visits;
* Ability to comply with all study requirements for the duration of the study, as outlined in the protocol, willing to submit to significant lifestyle changes that include diet, eating and exercise habits for the duration of the clinical study;
* Females of childbearing potential (FOCBP) must be willing to avoid pregnancy throughout the duration of the study, including follow-up, and must agree to the following:

  * have a negative serum pregnancy test as screening,
  * negative urine pregnancy test day of implant,
  * and inform the investigator immediately if the subject becomes pregnant;
* Willing to abstain from illegal drugs, including marijuana and tobacco (all forms) during study participation;
* Willing to limit alcohol consumption following the opinion of the Science Group of the European Alcohol and Health Forum of the European Commission;
* Has as stable concomitant medication regimen at the time of screening to mitigate drug induced weight fluctuations. A stable regimen is defined as 90 days without the introduction of or change in medication;
* Agrees to refrain from any type of reconstructive surgery/procedures that would affect body weight (such as abdominal lipoplasty or liposuction, mammoplasty, removal of excess skin or cool sculpting) during the follow-up period after the placement of the LGV.

Exclusion Criteria:

* Genetically-caused obesity, such as Prader-Willi syndrome; or any disease state know to affect weight status such as Cushing's syndrome, untreated sleep apnea, inadequately treated thyroid disease;
* History of chronic and/or ongoing clinically significant conditions or disorders of the gastrointestinal (GI) tract, i.e. Gastroparesis and Inflammatory Bowel Diseases such as Ulcerative Colitis and Crohn's disease;
* Any abnormal stenosis or obstruction of the GI tract;
* Significant acute and/or chronic active infection including H. pylori and urinary tract infection;
* History, or signs and/or symptoms of acid-peptic disease (APD) or gastric or duodenal ulcer;
* Diagnosis of portal hypertension, cirrhosis and esophageal varices;
* Presence of renal or liver disease defined as estimated Glomerular Filtration Rate (eGFR) < 45 ml/min/1.73 m2, ALT or AST > 2x upper limit normal (ULN) or total bilirubin >1.5x ULN;
* Previous stomach or bowel surgery;
* Previous bariatric procedure or device including, but not limited to, intragastric balloons within the past twelve months, sleeve gastrectomy, endoluminal suturing and restrictive bands;
* History of adhesive peritonitis;
* Presence of a hiatal hernia greater than 3 cm;
* History of bleeding disorders such as hemophilia;
* Unable to tolerate abstinence from blood thinners, such as warfarin, during the peri-operative period;
* Anemia defined as either: Hemoglobin (Hb) value for females of <11.0 g/dl, for males <12.0 g/dl;
* Abnormal blood cell indices deemed to be clinically significant;
* Diabetes requiring insulin at baseline (Type 1 or uncontrolled Type 2 defined as an HbA1c >12%) or a significant likelihood of requiring insulin treatment in the following 24 months;
* History or known allergies to silicone or similar materials;
* Participation in other investigational study protocols. If a subject has recently completed participation in another drug or device study, the subject must have exited that study at least 90 days prior to being enrolled in this study. If a subject screen failed prior to receiving study intervention the subject may participate in the study;
* Concomitant use of (or within 90 days of screening), or unwillingness to avoid any use of, weight loss medications, weight loss supplements, weight loss herbal preparations and/or participation in any non-study-related organized weight loss program (commercial or medical) at any time during the study;
* Undergoing chronic steroid or immunosuppressive therapy, defined as use of any oral and/or injectable steroid of any dose within 90 days of screening;
* Smoking cessation within two years of study entry;
* Major abdominal surgery (other than appendectomy, cholecystectomy);
* Significant traumatic injury to the abdomen within 90 days prior to enrollment;
* Subjects or immediate family members (e.g., biological parents, children, grandparents) with a known diagnosis or pre-existing symptoms of autoimmune connective tissue disease such as systemic lupus erythematosus or scleroderma;
* Current use of medications known to cause metabolic disturbances, such as the antipsychotic agents olanzapine, quetiapine, and type 2 diabetes medication thiazolidinedione (TZD);
* Chronic use of Non Steroid Anti-Inflammatory Drugs (NSAID) which is defined as daily use for greater than one month (daily low dose aspirin is acceptable);
* History or presence of malignancy such as cancer within the last five years with the exception of successfully treated non-melanoma skin cancer;
* Any condition that, in the opinion of the Investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
%Excess Weight Loss | 12 Months
  Demonstrate at least 30% excess weight loss (%EWL)
Rate of Related Serious Adverse Events | 12 Months
  Evaluate safety by device and procedure-related serious adverse events

SECONDARY OUTCOMES:
Rate of Related Serious Adverse Events | 24 months
  To evaluate the device and procedure-related serious adverse event rate
%Excess Weight Loss (EWL) | 24 Months
  To demonstrate the maintenance of at least 30% EWL
Percentage of Subjects With >=40% Excess Weight Loss (EWL) | 24 Months
  To demonstrate at least 40% EWL for at least 40% of subjects compared to baseline
Percentage of Subjects With >=50% Excess Weight Loss (EWL) | 24 Months
  To demonstrate at least 50% EWL for at least 35% of subjects compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dov Gal, Study Director — ReShape Lifesciences
Locations (1):
- Hospital universitario de Bellvitge, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No